CLINICAL TRIAL: NCT01606735
Title: A Multicenter, Randomized, Double-masked, Dose-ranging, Phase 2 Study to Evaluate the Efficacy and Safety of IBI-10090 for the Treatment of Inflammation Associated With Ocular Surgery
Brief Title: Efficacy and Safety of IBI-10090 in Ocular Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ICON Bioscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C11-01
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Inflammation Associated With Cataract Surgery
Keywords: cataract surgery; ocular inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Drug: IBI-10090
- Dose 2 (Experimental)
  Interventions: Drug: IBI-10090
- Dose 3 (Experimental)
  Interventions: Drug: IBI-10090

INTERVENTIONS:
Drug: IBI-10090 — dexamethasone

SUMMARY:
This study will test the efficacy and safety of IBI-10090 in the treatment of ocular inflammation after ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral cataract surgery

Exclusion Criteria:

* Ocular, topical, or oral corticosteroids within 7 days of Day 0

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Murahashi, MD, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Inland Eye Specialists, Hemet, California
  - California Eye Professionals, Temecula, California

RESULTS

PARTICIPANT FLOW:
Groups:
- 342 mcg; 517 mcg; 697 mcg: IBI-10090: dexamethasone
Period: Overall Study
Arm/Group | 342 mcg | 517 mcg | 697 mcg
Started | 58 | 56 | 58
Completed | 58 | 56 | 58
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 342 mcg | 517 mcg | 697 mcg | Total
Number analyzed (Participants) | 58 | 56 | 58 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.9) | 71.8 (71.8) | 70.1 (10) | 70.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 31 | 105
  Male | 23 | 17 | 27 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 2 | 2 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 5 | 7
  White | 50 | 51 | 45 | 146
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 58 | 56 | 58 | 172

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Count at Day 8 Post-Treatment
Description: This study will measure as its primary endpoint the anterior chamber cell count at Day 8 post-treatment. The proportion of patients with anterior chamber cell count = 0 at Day 8 for each dosage group will be compared.
Time Frame: 8 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with ACC clearing
Arm/Group | 342 mcg | 517 mcg | 697 mcg
Number analyzed (Participants) | 58 | 56 | 58
percentage of patients with ACC clearing | 50 [37.13 to 62.87] | 51.8 [38.7 to 64.87] | 60.3 [47.76 to 72.93]

ADVERSE EVENTS:
Arm/Group | 342 mcg | 517 mcg | 697 mcg
Serious Adverse Events (participants affected / at risk) | 6/58 | 2/56 | 3/58
Other Adverse Events (participants affected / at risk) | 2/58 | 2/56 | 1/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 342 mcg (N=58) | 517 mcg (N=56) | 697 mcg (N=58)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Corneal edema (Eye disorders) | 2 | 0 | 0
Corneal endothelial cell loss (Eye disorders) | 3 | 1 | 3
Endophthalmitis (Eye disorders) | 1 | 0 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 342 mcg (N=58) | 517 mcg (N=56) | 697 mcg (N=58)
Headache (Nervous system disorders) | 2 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information related to this study is considered confidential information belonging to Icon Bioscience, Inc. Data on the use of the study drug and results of all clinical and laboratory studies are considered private and confidential. None of the details, results, or other information for this study shall be published or made known to a third party without written consent from Icon Bioscience, Inc., except for disclosure to regulatory agencies if required by law.